CLINICAL TRIAL: NCT07303855
Title: Effectiveness of Goal-Directed Fluid Therapy Guided by Cardiac Index Versus Central Venous Pressure in Major Abdominal Surgery Patients in the ICU.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Sidharta K. Manggala, Principal investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-08-1273
Record Dates: First submitted 2025-11-29; First posted 2025-12-26 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Elective Major Abdominal Surgery
Keywords: cardiac index; central venous pressure; goal-directed fluid therapy; elective major abdominal surgery; postoperative fluid management; intensive care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Cardiac Index) (Experimental): During the first 6 hours postoperatively in the ICU, patients will receive fluid following a Goal-Directed Fluid Therapy (GDFT) protocol, with a target Cardiac Index of 2.5 to 4.0 L/min/m².
  Interventions: Procedure: Goal-Directed Fluid Therapy (GDFT)
- Group B (Central Venous Pressure) (Active Comparator): During the first 6 hours postoperatively in the ICU, patients will receive fluid following a Goal-Directed Fluid Therapy (GDFT) protocol, with a target Central Venous Pressure (CVP) of 8-12 mmHg.
  Interventions: Procedure: Goal-Directed Fluid Therapy (GDFT)

INTERVENTIONS:
Procedure: Goal-Directed Fluid Therapy (GDFT) — For the 6-hour intervention period, patients will receive fluid according to a Goal-Directed Fluid Therapy (GDFT) protocol. The treatment group will be managed to a target Cardiac Index of 2.5-4.0 L/min/m², while the control group will be managed to a target Central Venous Pressure (CVP) of 8-12 mmHg. All patients will receive a maintenance fluid volume of 25 mL/kg/24 hours, which will comprise the total volume from both parenteral fluids and enteral nutrition.

SUMMARY:
This study aims to compare two different methods for guiding intravenous (IV) fluid therapy in patients during their first 6 hours in the ICU after major abdominal surgery. The goal is to determine which method leads to a more optimal and precise amount of fluid administration. The objective is to compare the total fluid volumes administered when guided by Cardiac Index versus Central Venous Pressure, as well as mortality, length of stay, relaparotomy and reintubation in order to identify the more precise fluid management strategy for postoperative ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 to 65 years.
* Patients with a Body Mass Index (BMI) between 18 and 30 kg/m².
* Patients undergoing elective major abdominal surgery with a planned postoperative admission to the ICU.
* Patients with an American Society of Anesthesiologists (ASA) physical status classification of I to III.

Exclusion Criteria:

* Patients with pre-operative cardiovascular disorders (Coronary Artery Disease, or heart failure NYHA Class III and IV).
* Patients with severe renal impairment (Chronic Kidney Disease Stage V) with or without hemodialysis and fluid restrictions.
* Non-sinus cardiac rhythm.
* Pregnancy.
* Patients with right heart failure (patients with signs of congestion and symptoms of right heart failure accompanied by evidence of reduced right ventricular function, indicated by TAPSE < 17 mm).
* Patients with pulmonary hypertension (patients with echocardiographic suspicion of tricuspid regurgitation, tricuspid regurgitation velocity > 3.4 m/s, or mean pulmonary artery pressure > 20 mmHg from right heart catheterization).
* Patients with Acute Respiratory Distress Syndrome (ARDS) or patients requiring specialized ventilation modes.
* Patients who refuse to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Total Intravenous Fluid Volume in the ICU | From ICU enrollment until ICU discharge, up to 30 days
  The cumulative volume of intravenous fluids administered, recorded for both the initial 6-hour study period and the total ICU stay. Data will be obtained from ICU charts and recorded as a numerical value (mL).

SECONDARY OUTCOMES:
ICU Mortality | From ICU enrollment until ICU discharge, up to 30 days
ICU Length of Stay | From ICU enrollment until ICU discharge, up to 30 days
Relaparotomy | From ICU enrollment until ICU discharge, up to 30 days
  The occurrence of a relaparotomy procedure during the ICU stay, prior to step-down to a general ward.
Reintubation | From ICU enrollment until ICU discharge, up to 30 days
  The occurrence of a reintubation during the ICU stay, prior to step-down to a general ward.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No